CLINICAL TRIAL: NCT03668951
Title: Pharmacokinetic Study of Dexmedetomidine After Intra-Nasal and Buccal Dosing in Children
Acronym: DexPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-3034
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Heart Diseases
Keywords: Pediatric; Sedation; Dexmedetomidine
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Buccal DEX 2 mcg/kg (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia, placement of an endotracheal tube and an arterial line. Once these are accomplished, Dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine buccal
- Intranasal DEX 3 mcg/kg (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia, placement of an endotracheal tube and an arterial line. Once these are accomplished, Dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine Intranasal
- Intranasal DEX 4 mcg/kg (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia, placement of an endotracheal tube and an arterial line. Once these are accomplished, Dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine Intranasal

INTERVENTIONS:
Drug: Dexmedetomidine buccal — DEX 2 mcg/kg buccal
  Arms: Buccal DEX 2 mcg/kg
Drug: Dexmedetomidine Intranasal — DEX 3 mcg/kg intranasal
  Arms: Intranasal DEX 3 mcg/kg
Drug: Dexmedetomidine Intranasal — DEX 4 mcg/kg intranasal
  Arms: Intranasal DEX 4 mcg/kg

SUMMARY:
This research study is a continuation of a previous DEX PK study. It is examining the absorption of Dexmedetomidine (DEX) in the blood when given orally and as a nasal spray. This study will help us determine the best dosing amount for children undergoing sedation or anesthesia with DEX.

DETAILED DESCRIPTION:
The study will be a prospective study of plasma concentrations after intranasal or buccal DEX to determine the early pharmacokinetics and bioavailability of a single dose via nasal or oral administration.

Dexmedetomidine sedation is commonly used at Cincinnati Children's Medical Center and other pediatric institutions. This compound is typically delivered intravenously or intranasally for sedation in children with or without congenital heart disease. Intranasal DEX is very effective for sedation although it has significant variability in the onset and peak effect. Patient care will be improved if factors that determine this variability can be determined. Investigators will determine the important clinical variables of peak plasma DEX concentration (Tmax and Cmax) of intranasal and buccal DEX in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 - 48 months (inclusive) scheduled to receive anesthesia for elective cardiac surgery
* The subject must be a candidate to receive Dex as determined by one of the study cardiac anesthesiologists
* The attending cardiac anesthesiologists for the case and the Chief of Anesthesia Cardiac Anesthesia will concur with or veto this decision
* The subjects legally authorized representative has given written informed consent to participate in the study

Exclusion Criteria:

* Post-natal age less than 6 months
* The subject is allergic to or has had a contraindication to Dex
* Severely depressed ventricular function on preoperative echocardiogram
* The subject has a high risk of cardiac conduction system disease in the judgement of the attending anesthesiologist or cardiologist
* The subject has a hemodynamically significant aortic coarctation or other left heart outflow obstruction
* The subject has received digoxin, beta-adrenergic antagonist, or calcium channel antagonist on the day of surgery
* The subject has received Dex within 1 week of the study date
* Patients who are to receive intranasal Dex are excluded if they have nasal/respiratory symptoms, which in the opinion of the study anesthesiologist, may affect intranasal drug absorption

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum blood concentration level of Dex - Cmax | Blood samples will be drawn at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after Dex has been .
  Dex concentration will be measured in the blood to determine the time point with the maximum concentration (Cmax).
The amount of time that Dex is present at the maximum concentration - Tmax | Blood samples will be drawn at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after Dex has been .
  Dex concentration will be measured in the blood to determine the time point with the maximum concentration and how long that maximum concentration lasts.

SECONDARY OUTCOMES:
Area under the curve for Dex concentration levels | Blood samples will be drawn at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after Dex has been .
  Dex concentration will be measured in the blood samples.
Bioavailability of intranasal Dex relative to intravenous Dex for distribution - plasma concentration | Blood samples will be drawn at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after Dex has been .
  Data will also be analyzed using population modeling using nonlinear mixed effect modeling (NONMEM). Investigators will be measuring for approximately one half-life of Dex. This will allow us to estimate the important clinical parameter of relative bioavailability of intranasal vs intravenous Dex.
Bioavailability of IN Dex relative to intravenous Dex for elimination - plasma concentration. | Blood samples will be drawn at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after Dex has been .
  Data will also be analyzed using population modeling using nonlinear mixed effect modeling (NONMEM). Investigators will be measuring for approximately one half-life of Dex. This will allow us to estimate the important clinical parameter of relative bioavailability of intranasal vs intravenous Dex.
Adverse events associated with Dex administration | Participants will be followed until cardiopulmonary bypass, an expected duration of 2 hours.
  Heart rate will be recorded by clinical staff prior to the procedure and continuously during the procedure. The heart rate during the time of study blood collection will be compared to the baseline vitals to determine is any adverse events occurred.
Systolic and diastolic blood pressure with Dex administration | Participants will be followed until cardiopulmonary bypass, an expected duration of 2 hours.
  Systolic and diastolic blood pressure will be recorded by clinical staff prior to the procedure and continuously during the procedure. The systolic and diastolic blood pressure during the time of study blood collection will be compared to the baseline blood pressure to determine is any adverse events occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Pratap, MA,MB BChir,MRCPCH,FRCA, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Joanna Paquin, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No